CLINICAL TRIAL: NCT02000700
Title: Open-Label, Multicenter, Multiple Oral Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Canagliflozin in Older Children and Adolescents ≥10 to <18 Years of Age With Type 2 Diabetes Mellitus and Currently on a Stable Dose of Metformin
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Canagliflozin in Older Children and Adolescents With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103045; 28431754DIA1055 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Canagliflozin; JNJ-28431754; Pharmacokinetics; Pharmacodynamics; Children; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

ARMS (2):
- Canagliflozin (Dose Group 1) (Experimental): Participants will receive 100 mg (as 1 x 100-mg tablet) of canagliflozin daily for 14 days.
  Interventions: Drug: Canagliflozin 100 mg; Drug: Placebo
- Canagliflozin (Dose Group 2) (Experimental): Participants will be enrolled into Dose Group 2 to receive either 50 mg (as 1 x 50-mg tablet) or 300 mg (as 1 x 300-mg tablet) of canagliflozin daily for 14 days.
  Interventions: Drug: Canagliflozin 50 mg; Drug: Canagliflozin 300 mg; Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 100 mg — One 100-mg tablet of canagliflozin orally administered daily for 14 days.
  Arms: Canagliflozin (Dose Group 1)
Drug: Canagliflozin 50 mg — One 50-mg tablet of canagliflozin orally administered daily for 14 days.
  Arms: Canagliflozin (Dose Group 2)
Drug: Canagliflozin 300 mg — One 300-mg tablet of canagliflozin orally administered daily for 14 days.
  Arms: Canagliflozin (Dose Group 2)
Drug: Placebo — One matching placebo tablet orally administered at baseline phase.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (blood levels) and pharmacodynamics (the action or effects a drug has on the body) of canagliflozin in children and adolescents with type 2 diabetes mellitus aged 10 to 17 years (inclusive). Other purposes are to investigate safety and assess the ease of swallowing the tablets.

DETAILED DESCRIPTION:
The participants who meet the eligibility criteria, will receive a single dose of placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) and this will be followed by baseline 24 hour pharmacodynamic assessments. On the next morning participants will receive the first canagliflozin dose and will be discharged home to continue canagliflozin treatment for 13 additional days. There will be 2 treatment groups (8 participants in each): the first group will receive canagliflozin 100 mg daily, the second group will receive either canagliflozin 300 mg or canagliflozin 50 mg daily. The canagliflozin dose for the second treatment group will be determined after the sponsor has evaluated the results from the first 5 participants. On day 14 of treatment the participants will be admitted again for 24 hour pharmacokinetic and pharmacodynamics assessments. The participants will continue to take their normal dose and schedule of metformin during the entire study. The total duration of the study is approximately 50 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus
* Be on a stable regimen of metformin immediate release (IR) monotherapy of at least 1,000 mg/day for at least 8 weeks before screening
* Able to swallow whole tablets
* Absence of pancreatic autoimmunity
* Participants and their caregivers must agree to perform the fasting fingerstick glucose self-monitoring during the study

Exclusion Criteria:

* History of Type 1 diabetes mellitus
* History of maturity onset diabetes of the young (MODY) and any secondary form of diabetes
* Current clinically significant medical illness e.g., significant pulmonary disease, renal or hepatic insufficiency, uncontrolled thyroid disease
* Systolic or diastolic blood pressure outside the range considered normal for the participant sex, age and height
* For females, participants will be excluded if pregnant

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin following multiple oral doses of canagliflozin | From Days 14 to 17
  Plasma concentrations of canagliflozin are used to evaluate how long canagliflozin stays in the body.

SECONDARY OUTCOMES:
Plasma glucose concentration following multiple oral doses of canagliflozin | From Days -1 to 1, and from Days 14 to 15
  Plasma glucose is equal to the amount of glucose in the plasma at the defined time points.
Urine glucose excretion following multiple oral doses of canagliflozin | From Days -1 to 1, and from Days 14 to 15
  Urine glucose excretion is equal to the amount of glucose excreted into the urine over defined time intervals.
Renal threshold for glucose excretion following multiple oral doses of canagliflozin | From Days -1 to 1, and from Days 14 to 15
  Renal threshold is defined as the plasma glucose concentration above which glucose is excreted in the urine.
Acceptability of the canagliflozin tablet | Day 14
  A questionnaire containing 5 questions about the acceptability of the tablet (taste, smell, swallowability, residual mouth taste, and overall feeling) will be administered to the participants at the end of the treatment phase. Each question is rated using a 5 or 6-point scale. The scales comprise the following outcomes: very negative, negative, neutral, positive, and very positive. Results will be summarized descriptively.
Number of participants with adverse events as a measure of safety and tolerability | Approximately 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- United States (13):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Indianapolis, Indiana
  - Lenexa, Kansas
  - Baltimore, Maryland
  - Kansas City, Missouri
  - Toledo, Ohio
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Salt Lake City, Utah
- Brazil (4):
  - Campinas
  - Curitiba
  - Ribeirão Preto
  - São Paulo

REFERENCES:
- See also: Open-Label, Multicenter, Multiple Oral Dose Study to Evaluate Pharmacokinetics, Pharmacodynamics and Safety of Canagliflozin in Older Children and Adolescents ≥10 to <18 years' age with Type 2 Diabetes Mellitus and Currently on a Stable Dose of Metformin — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=5713&filename=CR103045_CSR.pdf